CLINICAL TRIAL: NCT01359891
Title: Clinical Evaluation of Novel Biomarkers for Diagnosis, Therapy- Monitoring and Prognosis of Outcome in Patients With Septicemia
Brief Title: Clinical Evaluation of Novel Biomarkers in Patients With Septicemia
Acronym: NOBIS
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Robert Krause, MD, ao.Univ.Prof.Dr, Medical University of Graz
Other Study IDs: 21-469
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Sepsis; Bacteremia; Fungemia
MeSH Terms: conditions — Sepsis; Bacteremia; Fungemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Left over EDTA-whole blood samples will be used for both, the Presage™ST2 assay and the suPARnostic™ assay except for the additional EDTA-whole blood samples taken on day 1 and 2 of study enrollment being only tested for sST2.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cohort 1: All patients >18 years admitted to the University Hospital Graz, Austria, with positive blood cultures tested in the Microbiology Laboratory, Department of Internal Medicine, Medical University Graz, or the Institute for Hygiene, Microbiology and Environmental Medicine, Medical University Graz, are screened for study inclusion. Patients eligible for the study have to have Staphylococcus aureus, Escherichia coli, Pseudomonas aeruginosa, Enterococcus faecium, Enterococcus faecalis, Streptococcus pneumoniae, Klebsiella pneumoniae or medically relevant fungi / viral pathogens identified as causative pathogen.
  The estimated total number of patients included in this first study cohort will be 500.
- Cohort 2: All patients >18 years admitted to the University Hospital Graz, Austria, will be screened for study inclusion if the attending emergency department physicians on the very first visit suspects bacteremia/fungemia/sepsis and consecutively orders blood cultures. Patients will be included in this second cohort if these initially taken blood culture turns positive (n=200) or stays negative (n=50) at the Microbiology Laboratory, Department of Internal Medicine, Medical University Graz. As soon as the number of 50 is reached for the control group enrollment will be stopped for this group.
  As soon as the proposed number of 250 patients is reached enrolment for this second cohort will be stopped. Patients enrolled in cohort 2 may also be consecutively enrolled in cohort 1.
- Validation Cohort: To verify the employed Presage™ST2 assay established in our study laboratory for its intended use, a total number of 70 left over plasma samples obtained from septic patients which have prior been tested for sST2 with the same assay at the Department of Laboratory Medicine, Barmherzige Brueder Linz, Austria, will be retested. This cohort therefore serves as a validation cohort.

SUMMARY:
The protein ST2 is a member of the interleukin-1 receptor family. Blood concentrations of the soluble isoform of ST2 (sST2) are increased in inflammatory and heart diseases and are considered a prognostic marker in both. The Presage™ST2 assay was recently shown to meet the needs of quality specifications of laboratory medicine. Soluble urokinase plasminogen activator receptor (suPAR) levels reflect inflammation and elevated suPAR levels are found in several infectious diseases and cancer. Both sST2 and suPAR have recently been introduced as sensitive biomarkers for patients with septicemia. Both may be promising or even superior alternatives to currently established sepsis markers leading to an improvement of outcome in patients with septicemia. However, a clinical study which clarifies kinetics of values over time/possible correlation with causative pathogen/progress/deterioration of septic patients is urgently needed before these biomarkers can be established in clinical routine.

Primary study objectives To clinically evaluate sST2 and suPAR in patients with bacteremia /septicemia. To correlate results with causative bacterial organisms, response to or failure of antiinfective treatment, severity of clinical status as well as outcome.

To study the kinetics of the test results and to correlate the sST2/suPAR results with other well established infection markers (e.g. C-reactive protein, procalcitonin, blood counts).

Natural endpoints of the study will be patient's death or complete recovery.

This is an explorative study. To meet the objectives both novel biomarkers will be clinically evaluated in a cohort of 500 in-patients with septicemia at the University Hospital Graz. Starting the day a patient's blood culture turned positive the investigators will collect samples every 12h within the first two days and then every 24h.Measurement of sST2 and suPAR values will be done retrospectively. To analyze clinical sensitivity/specificity of the novel biomarkers sST2 and suPAR as prognostic factors for development of bacteremia/septicemia, a second cohort consisting of 250 in-patients will be investigated in a longitudinal matter. Patients without a previous positive blood culture test during the current episode of disease for which blood cultures are ordered by a physician will be included and sST2 and suPAR levels will be determined from samples taken simultaneously with this first blood cultures.

DETAILED DESCRIPTION:
The two most common causative pathogens of septicemia (Escherichia coli and Staphylococcus aureus) as well as cases of fungemia (Candida spp., Aspergillus spp., and others) will be included in the first study group. At our hospital the estimated yearly cases of bacteremia/fungemia (230 for Escherichia coli, 150 for Staphylococcus aureus, and 50 for fungi) will be included in the first study group. Furthermore, the two biomarkers will be determined in 70 cases of septicemia with other bacterial pathogens and sepsis due to viral pathogens or viremia for evaluation of further clinical impact of these two biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years

Exclusion Criteria:

* Patients < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18years with suspected / proven bacteremia/septicaemia admitted to the medical university hospital Graz, Austria
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2010-11; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
prognostic value of biomarkers in bacteremia | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hoenigl, MD, Principal Investigator — Medical University of Graz; Robert Krause, MD, Principal Investigator — Medical University of Graz; Reinhard R Raggam, MD, Principal Investigator — Medical University Hospital Graz
Locations (1):
- Medical University Hospital of Graz, Graz, Styria, Austria